CLINICAL TRIAL: NCT03172559
Title: A Multi-Center Randomized Controlled Trial Comparing Stereotactic Body Radiotherapy as a "Bridge" Prior to Liver Transplant for Hepatocellular Carcinoma Versus no Intervention in Patients Not Eligible to Transarterial Chemoembolization or Ablation
Brief Title: Radiotherapy Versus no Intervention in Adult Patients With Hepatocellular Carcinoma Not Eligible for Transarterial Chemoembolization or Ablation Prior to Liver Transplant (RADBRI)
Acronym: RADBRI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decided not to pursue the study due to other competing studies.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-5329
Record Dates: First submitted 2017-04-05; First posted 2017-06-01 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Stereotactic body radiotherapy; SBRT; Radiotherapy; Bridging therapy; Transplant
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Explanatory, multicenter, open label, 2-arm parallel group superiority randomized trial with stratification by center and blood group, random permuted blocks (lengths of 4 or 6) and balanced allocation (1:1).
Who Masked: Outcomes Assessor
Masking Description: The data manager uploading the data into a database and the statistician analyzing the data will be blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic body radiotherapy (Experimental): Stereotactic body radiotherapy (SBRT) treatment will be individualized with the dose based on baseline liver function, effective liver volume irradiated and proximity to other normal tissues. The recommended dose will be 30 gray (Gy) in 5 fractions. The treatment will be administered in 5 alternative days. Patients will come every other day to the hospital to be treated and will not need to be admitted. Patients will not receive further SBRT on the treated tumor.
  Interventions: Radiation: Stereotactic body radiotherapy
- No intervention (No Intervention): Follow-up will be carried out every 3 months and a computed tomography (CT) scan of the chest and abdomen or an magnetic resonance imaging (MRI), and blood work with liver function test and alpha-fetoprotein (AFP) value will be done until the patient is transplanted or drops-out of the waiting list.

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — The recommended dose will be 30 Gy in 5 fractions. The treatment will be administered in 5 alternative days and will be individualized with the dose based on baseline liver function, effective liver volume irradiated and proximity to other normal tissues.
  Other Names: SBRT
  Arms: Stereotactic body radiotherapy

SUMMARY:
Liver transplantation (LT) represents the best treatment for patients with selected, early stage hepatocellular carcinoma (HCC). Due to the gap between the number of patients on the waiting list and the available donors, patients with HCC wait ~1 year to be transplanted. While waiting, 25-30% of patients need to come off the transplant list due to tumor progression beyond transplant criteria (extrahepatic disease, vascular invasion or increase in tumor burden beyond enlistment criteria). To try to avoid this progression, patients are treated while waiting with "bridging therapies", mainly transarterial chemoembolization (TACE) and ablation. Around 30% of patients are not eligible for these treatments (.e.g. due to poor liver function). Stereotactic body radiotherapy (SBRT) has been shown to be an effective treatment for advanced HCC in primarily small, single institutional studies and its safety has been reported in cirrhotics. SBRT could be used in patients not eligible to TACE or ablation as a bridge to LT reducing the risk of progression in the waiting list. This study will evaluate if patients with liver cirrhosis and HCC benefit from receiving SBRT while awaiting LT. Patients will be randomized to a treatment arm where they will receive SBRT as a bridge therapy or to a no intervention arm. Outcomes prior and post to transplant will be performed to evaluate the differences between both arms: proportion of patients that do not drop-out of the list (are transplanted), liver decompensation while waiting, perioperative measures in those that are transplanted, time to transplant or drop-out, overall survival, disease-free survival in those that are transplanted in a population of about 330 patients across all sites.

DETAILED DESCRIPTION:
The RADBRI trial is designed as an explanatory, multicenter, open-label, 2-arm parallel group superiority randomized trial with stratification by center and blood group, random permuted blocks (lengths of 4 or 6) and balanced allocation (1:1) conducted in 8 centers across the world. Including a population of adult patients with hepatocellular carcinoma (HCC) included in the waiting list for a liver transplant (LT) that are not eligible for transarterial chemoembolization (TACE) or ablation as a bridge to transplant but are eligible to stereotactic body radiotherapy (SBRT). Participants will be randomly assigned to either no intervention or SBRT with a 1:1 allocation as per an online, central randomization service (Sealed Envelope™) and stratified by site and by blood type (ABO type) using random permuted blocks (lengths 4 or 6). Aiming for a total sample of 332 (166 per group). Patients will be followed for 18 months until drop-out from waiting list or LT. A computed tomography (CT) or magnetic resonance imaging (MRI) and alpha-fetoprotein (AFP) level will be performed every 3 months while waiting. In those that get transplanted, follow-up will be carried out for additional 36 months (every 3 months for the first 2 years and every 6 months thereafter).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Patient has been included in the waiting list to receive a Liver Transplant (LT)
* Radiological confirmation of Hepatocellular carcinoma (HCC) according to American Association for the Study of Liver Diseases (AASLD) guidelines
* Tumor burden at randomization within a total tumor volume (TTV) ≤115 cm3 and serum alpha-fetoprotein (AFP) ≤400 ng/mL
* Patient not eligible to bridging therapy with Transarterial Chemoembolization (TACE) and/or ablation.
* Child-Pugh score ≤B9
* Calculated Model of End Stage Liver disease (MELD) score ≤20
* Eligible to Stereotactic body radiotherapy (SBRT): >40% of liver parenchyma can be spared from radiation and all tumors can be targeted
* No previous treatment of the tumor
* Absence of extra-hepatic disease or vascular invasion on imaging
* Able and willing to provide consent

Exclusion Criteria:

* Patient with HCC not candidate to receive a LT
* Patient is eligible to TACE or ablation as a bridge to LT
* Patient is not eligible to SBRT
* Previous bridging therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Difference between the two treatment arms in the proportion of participants that get to be transplanted (do not drop-out from the waiting list due to tumor progression). | 5 years
  Treatment success is defined as being transplanted. Treatment failure is defined as dropping off the waiting list for any cause (tumor progression or liver decompensation)

SECONDARY OUTCOMES:
Difference between the two arms in liver decompensation while waiting | 5 years
  Defined as an increase in the Child-Pugh score measured in each follow-up visit while the patient is in the waiting list will be compared between patients in each arm
Difference between the two arms in perioperative measures | 5 years
  Proportion of patients with major complications measured in the first 90 days post Liver Transplant
Difference between the two arms in time to transplant or drop-out | 5 years
  Time to event (drop-out or transplant) between both groups
Difference between the two arms in overall survival | 5 years
  Time-to-event between both groups. This comparison will be done from the time of randomization and from the time of Liver Transplant (LT) in those that get transplanted. Causes of death after transplant will be collected and compared between groups.
Difference between the two arms in overall survival | 5 years
  Time-to-event between both groups. This comparison will be done from the time of randomization and from the time of Liver Transplant (LT) in those that get transplanted. We will assess the effect of Stereotactic body radiotherapy (SBRT) post LT and this will be used a hypothesis generating information for future trials
Difference between the two arms in disease-free survival | 5 years
  Time-to-event between both groups. Tumor recurrence (new Hepatocellular carcinoma after liver transplant) and patterns of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, Principal Investigator — University Health Network, Toronto; Laura Dawson, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No